CLINICAL TRIAL: NCT06228872
Title: Direct Current Transcranial Stimulation as Cognitive Rehabilitation Therapy in Post-Traumatic Brain Injury Patients.
Brief Title: "Cognitive Rehabilitation With Direct Current Transcranial Stimulation in Post-Traumatic Brain Injury Patients"
Acronym: tDCS-TEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mutual de Seguridad Hospital Clinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Resolution number 340
Record Dates: First submitted 2023-07-06; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Traumatic Brain Injury; Cognitive Impairment
Keywords: Transcranial direct current stimulation (tDCS); Computerized cognitive training (CCT); Traumatic brain injury (TBI); Cognitive Impairment
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The study is a prospective, controlled, double-blind, randomized clinical trial in collaboration with the University of Chile. It includes patients with moderate cognitive impairment due to moderate-to-severe traumatic brain injury lasting over 6 months. Participants will be randomly assigned to the experimental or control group. The intervention involves computerized cognitive training (CCT) through a mobile app and daily self-administered transcranial direct current stimulation (tDCS) therapy to the prefrontal dorsolateral cortex (PFDL) for one month. Prior to the intervention, a training session will instruct patients on device use and adverse effects monitoring. Neuropsychological evaluations will be conducted at baseline (T0), immediately after the last session (T1), and one month later (T2). This trial aims to assess the efficacy of combined CCT and tDCS for cognitive impairment in TBI patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this trial, masking will ensure blinding of interventions:
  Participant: They will be unaware of receiving active tDCS therapy or sham intervention. A remote-controlled mobile app will facilitate this.
  Investigator: They will be masked, not knowing the assigned interventions. This minimizes bias in data collection and analysis.
  Outcomes Assessor: They will be masked to assigned interventions, ensuring objective and unbiased outcome assessment.
  Implementing masking ensures that participants, care providers, investigators, and outcomes assessors remain unaware of the intervention received, maintaining trial integrity and validity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants will receive Computerized Cognitive Training and anodal tDCS daily for one month. Stimulation will consist of 20 min of anodal 2mA tDCS stimulation over the DLPFC, followed by 15 min of computerized cognitive training.
  Interventions: Device: Cognitive Computerized Training (CCT) plus Anodic transcranial Direct Current Stimulation (tDCS)
- Control Group (Sham Comparator): Participants will receive Computerized Cognitive Training and sham tDCS daily for one month. Sham stimulation will consist of 60 seconds of anodal 2mA tDCS stimulation over the DLPFC, followed by 19 mins of no current delivery. The same 15 min of computerized cognitive training will be provided after the end of the Sham Stimulation.
  Interventions: Device: Cognitive Computerized Training (CCT) plus sham transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Cognitive Computerized Training (CCT) plus Anodic transcranial Direct Current Stimulation (tDCS) — Computerized Cognitive Training (15 min) + Anodal tDCS over DLPFC (20 min) daily for 1 month
  Arms: Experimental Group
Device: Cognitive Computerized Training (CCT) plus sham transcranial Direct Current Stimulation (tDCS) — Computerized Cognitive Training (15 min) + Sham tDCS over DLPFC (20 min) daily for 1 month
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to investigate the impact of daily self-administered transcranial direct current stimulation (tDCS) therapy on the cognitive function of individuals with moderate to severe cognitive impairment resulting from a traumatic brain injury (TBI). The study aims to answer the following questions:

Does daily self-administered tDCS therapy, when combined with computerized cognitive training (CCT), improve cognitive function in TBI patients? Is CCT+tDCS with anodic stimulation more effective than CCT+tDCS with simulated stimulation in enhancing immediate and one-month post-treatment cognitive function? Does CCT+tDCS with anodic stimulation lead to better functionality immediately and one month after treatment compared to CCT+tDCS with simulated stimulation? Does CCT+tDCS with anodic stimulation have a positive impact on mood improvement immediately and one month after treatment compared to CCT+tDCS with simulated stimulation? Participants in the study will engage in CCT through a smartphone or tablet application and self-administer tDCS therapy for 20 minutes each day for a duration of one month. The tDCS therapy will involve applying a 2 mA anodic current to the prefrontal dorsolateral cortex (PFDL). Prior to the intervention, patients or their caregivers will receive training on the proper and safe usage of the tDCS device. Cognitive function, mood, and functionality will be evaluated before and after the intervention using appropriate measurement scales.

The outcomes of this clinical trial have the potential to identify an effective and accessible therapeutic approach to enhance cognitive function in individuals with moderate to severe TBI. The combination of tDCS therapy with CCT offers an appealing and feasible treatment strategy for these patients, particularly when conducted in a home setting. The findings from this study will guide future clinical trials in the field of cognitive rehabilitation for TBI patients. Researchers will compare active tDCS with sham tDCS to determine if there are differences in the primary outcomes mentioned.

DETAILED DESCRIPTION:
Introduction: Transcranial direct current stimulation (tDCS) is a non-invasive neuromodulation technique that can modulate neuronal excitability and enhance neuroplasticity. On the other hand, computerized cognitive training (CCT) therapy uses computers to improve cognitive domains through repeated practice of theoretically-driven skills and strategies. So far, the isolated use of tDCS and its combination with CCT have been explored in the cognitive recovery of patients with traumatic brain injury (TBI), yielding promising results. However, none of the studies to date have investigated the use of a self-administered therapy (by the patient and/or caregiver) that combines both interventions at home. The objective of this clinical trial is to evaluate the effect of daily self-administered tDCS therapy on cognitive function in patients with moderate-to-severe TBI-associated cognitive impairment.

Methodology: A prospective, controlled, double-blind, randomized clinical trial is proposed. The intervention will consist of (i) CCT delivered through a smartphone or tablet application and (ii) the application of 2 mA tDCS therapy (20 minutes of anodic current for the experimental group and 60 seconds for the control group) to the prefrontal dorsolateral cortex (PFDL) daily for one month, self-administered by the patient. Prior to the intervention, a training session will be conducted to instruct the patient (or caregiver) on the correct and safe use of the device. The primary outcomes will be cognitive function, mood, and functionality, measured before and after the intervention using appropriate scales.

Discussion: The results of this clinical trial could contribute to the identification of an effective and accessible therapeutic method to improve cognitive function in patients with moderate-to-severe TBI. The combination of tDCS therapy with CCT may offer an attractive and feasible therapeutic strategy for these patients, particularly when performed at home. The findings of this study may be useful in guiding future clinical trials in the field of cognitive rehabilitation in TBI patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years.
* Moderate to severe traumatic brain injury (TBI) according to classification 58 (see Table 3) with a duration of 6 to 12 months.
* Minimum of 8 years of education (completed basic education with literacy skills).
* Meeting diagnostic criteria (see Table 3) for mild or major cognitive impairment according to the Diagnostic and Statistical Manual of Mental Disorders (DSM).
* Capacity to make decisions and understand relevant information regarding participation in a clinical trial, assessed using the MacArthur Competence Assessment Tool for Clinical Research (MacCAT-CR) 60.
* Inclusion of patients with chronic TBI (defined for this study as more than 6 months of duration) based on the proposed mechanism of chronic TBI involving decreased cerebral neuroplasticity, leading to long-term cognitive dysfunction and functional limitations 62. Transcranial Direct Current Stimulation (tDCS) has shown effectiveness in enhancing neuroplasticity in various neurological and psychiatric conditions 63.

Exclusion Criteria:

* History of cognitive impairment unrelated to post-traumatic causes (for which the patient is being treated at Mutual de Seguridad).
* History of epileptic seizures.
* Pre-existing neuropsychiatric disorders.
* Presence of metallic objects in the body such as aneurysm implants, hemostatic clips, implanted electrodes, and electrical devices like pacemakers.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Executive Cognitive function (Working Memory) | Baseline (T0), immediate post-treatment (T1), and one month post-treatment (T2).
  Measurement of working memory using Digit Span forward and backward.
Executive Cognitive Function | Baseline (T0), immediate post-treatment (T1), and one month post-treatment (T2).
  Assessment of general executive cognitive function using Ineco Frontal Screening (IFS) evaluation.

SECONDARY OUTCOMES:
Mood | Baseline (T0), immediate post-treatment (T1), and one month post-treatment (T2).
  Assessment of mood using the Structured Clinical Interview for Depression (SCID) to detect depressive symptoms.
Functional Independence | Baseline (T0), immediate post-treatment (T1), and one month post-treatment (T2).
  Evaluation of functional independence using the Functional Independence Measure (FIM) associated with the Functional Assessment Measure (FAM). FIM assesses independence in various domains of activities of daily living, while FAM is used to measure functionality and performance in daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Matamala Capponi, MD, Principal Investigator — Associated Professor of the University of Chile
Locations (1):
- Hospital de Mutual de Seguridad, Santiago, Metropolitan Region, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deidda G, Bozarth IF, Cancedda L. Modulation of GABAergic transmission in development and neurodevelopmental disorders: investigating physiology and pathology to gain therapeutic perspectives. Front Cell Neurosci. 2014 May 22;8:119. doi: 10.3389/fncel.2014.00119. eCollection 2014. PMID 24904277
- [Background] Fernandez E, Bringas ML, Salazar S, Rodriguez D, Garcia ME, Torres M. Clinical impact of RehaCom software for cognitive rehabilitation of patients with acquired brain injury. MEDICC Rev. 2012 Oct;14(4):32-5. doi: 10.37757/MR2012V14.N4.8. PMID 23154316
- [Background] Kang EK, Kim DY, Paik NJ. Transcranial direct current stimulation of the left prefrontal cortex improves attention in patients with traumatic brain injury: a pilot study. J Rehabil Med. 2012 Apr;44(4):346-50. doi: 10.2340/16501977-0947. PMID 22434324
- [Background] Hyder AA, Wunderlich CA, Puvanachandra P, Gururaj G, Kobusingye OC. The impact of traumatic brain injuries: a global perspective. NeuroRehabilitation. 2007;22(5):341-53. PMID 18162698
- [Background] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411
- [Background] Dikmen S, Machamer J, Fann JR, Temkin NR. Rates of symptom reporting following traumatic brain injury. J Int Neuropsychol Soc. 2010 May;16(3):401-11. doi: 10.1017/S1355617710000196. Epub 2010 Mar 1. PMID 20188017
- [Background] Jaeggi SM, Seewer R, Nirkko AC, Eckstein D, Schroth G, Groner R, Gutbrod K. Does excessive memory load attenuate activation in the prefrontal cortex? Load-dependent processing in single and dual tasks: functional magnetic resonance imaging study. Neuroimage. 2003 Jun;19(2 Pt 1):210-25. doi: 10.1016/s1053-8119(03)00098-3. PMID 12814572
- [Background] Bolognini N, Pascual-Leone A, Fregni F. Using non-invasive brain stimulation to augment motor training-induced plasticity. J Neuroeng Rehabil. 2009 Mar 17;6:8. doi: 10.1186/1743-0003-6-8. PMID 19292910
- [Background] Lesniak M, Polanowska K, Seniow J, Czlonkowska A. Effects of repeated anodal tDCS coupled with cognitive training for patients with severe traumatic brain injury: a pilot randomized controlled trial. J Head Trauma Rehabil. 2014 May-Jun;29(3):E20-9. doi: 10.1097/HTR.0b013e318292a4c2. PMID 23756431
- [Background] Sozda CN, Muir JJ, Springer US, Partovi D, Cole MA. Differential learning and memory performance in OEF/OIF veterans for verbal and visual material. Neuropsychology. 2014 May;28(3):347-352. doi: 10.1037/neu0000043. Epub 2013 Nov 18. PMID 24245926
- [Background] Stagg CJ, Best JG, Stephenson MC, O'Shea J, Wylezinska M, Kincses ZT, Morris PG, Matthews PM, Johansen-Berg H. Polarity-sensitive modulation of cortical neurotransmitters by transcranial stimulation. J Neurosci. 2009 Apr 22;29(16):5202-6. doi: 10.1523/JNEUROSCI.4432-08.2009. PMID 19386916
- [Background] Jak AJ, Seelye AM, Jurick SM. Crosswords to computers: a critical review of popular approaches to cognitive enhancement. Neuropsychol Rev. 2013 Mar;23(1):13-26. doi: 10.1007/s11065-013-9226-5. Epub 2013 Feb 20. PMID 23423553
- [Background] Kueider AM, Parisi JM, Gross AL, Rebok GW. Computerized cognitive training with older adults: a systematic review. PLoS One. 2012;7(7):e40588. doi: 10.1371/journal.pone.0040588. Epub 2012 Jul 11. PMID 22792378
- [Background] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Background] Russo C, Souza Carneiro MI, Bolognini N, Fregni F. Safety Review of Transcranial Direct Current Stimulation in Stroke. Neuromodulation. 2017 Apr;20(3):215-222. doi: 10.1111/ner.12574. Epub 2017 Feb 21. PMID 28220641
- [Background] Ulam F, Shelton C, Richards L, Davis L, Hunter B, Fregni F, Higgins K. Cumulative effects of transcranial direct current stimulation on EEG oscillations and attention/working memory during subacute neurorehabilitation of traumatic brain injury. Clin Neurophysiol. 2015 Mar;126(3):486-96. doi: 10.1016/j.clinph.2014.05.015. Epub 2014 Jun 2. PMID 24947595
- [Background] Sacco K, Galetto V, Dimitri D, Geda E, Perotti F, Zettin M, Geminiani GC. Concomitant Use of Transcranial Direct Current Stimulation and Computer-Assisted Training for the Rehabilitation of Attention in Traumatic Brain Injured Patients: Behavioral and Neuroimaging Results. Front Behav Neurosci. 2016 Mar 31;10:57. doi: 10.3389/fnbeh.2016.00057. eCollection 2016. PMID 27065823
- [Background] Quinn DK, Upston J, Jones T, Brandt E, Story-Remer J, Fratzke V, Wilson JK, Rieger R, Hunter MA, Gill D, Richardson JD, Campbell R, Clark VP, Yeo RA, Shuttleworth CW, Mayer AR. Cerebral Perfusion Effects of Cognitive Training and Transcranial Direct Current Stimulation in Mild-Moderate TBI. Front Neurol. 2020 Oct 7;11:545174. doi: 10.3389/fneur.2020.545174. eCollection 2020. PMID 33117255
- [Background] Eilam-Stock T, George A, Charvet LE. Cognitive Telerehabilitation with Transcranial Direct Current Stimulation Improves Cognitive and Emotional Functioning Following a Traumatic Brain Injury: A Case Study. Arch Clin Neuropsychol. 2021 Apr 21;36(3):442-453. doi: 10.1093/arclin/acaa059. PMID 33885138
- [Background] Fawcett J. Molecular control of brain plasticity and repair. Prog Brain Res. 2009;175:501-9. doi: 10.1016/S0079-6123(09)17534-9. PMID 19660677
- [Background] Demirtas-Tatlidede A, Vahabzadeh-Hagh AM, Bernabeu M, Tormos JM, Pascual-Leone A. Noninvasive brain stimulation in traumatic brain injury. J Head Trauma Rehabil. 2012 Jul-Aug;27(4):274-92. doi: 10.1097/HTR.0b013e318217df55. PMID 21691215
- [Background] Li S, Zaninotto AL, Neville IS, Paiva WS, Nunn D, Fregni F. Clinical utility of brain stimulation modalities following traumatic brain injury: current evidence. Neuropsychiatr Dis Treat. 2015 Jun 30;11:1573-86. doi: 10.2147/NDT.S65816. eCollection 2015. PMID 26170670
- [Background] Capizzi A, Woo J, Verduzco-Gutierrez M. Traumatic Brain Injury: An Overview of Epidemiology, Pathophysiology, and Medical Management. Med Clin North Am. 2020 Mar;104(2):213-238. doi: 10.1016/j.mcna.2019.11.001. PMID 32035565
- [Background] McInnes K, Friesen CL, MacKenzie DE, Westwood DA, Boe SG. Mild Traumatic Brain Injury (mTBI) and chronic cognitive impairment: A scoping review. PLoS One. 2017 Apr 11;12(4):e0174847. doi: 10.1371/journal.pone.0174847. eCollection 2017. PMID 28399158
- [Background] Motes MA, Spence JS, Yeatman K, Jones PM, Lutrell M, O'Hair R, Shakal S, DeLaRosa BL, To W, Vanneste S, Kraut MA, Hart J , Jr. High-Definition Transcranial Direct Current Stimulation to Improve Verbal Retrieval Deficits in Chronic Traumatic Brain Injury. J Neurotrauma. 2020 Jan 1;37(1):170-177. doi: 10.1089/neu.2018.6331. Epub 2019 Sep 3. PMID 31354040